CLINICAL TRIAL: NCT04444674
Title: An Adaptive Phase I/II Randomized Placebo-controlled Trial to Determine Safety, Immunogenicity and Efficacy of Non-replicating ChAdOx1 SARS-CoV-2 Vaccine in South African Adults Living Without HIV; and Safety and Immunogenicity in Adults Living With HIV
Brief Title: COVID-19 Vaccine (ChAdOx1 nCoV-19) Trial in South African Adults With and Without HIV-infection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council, South Africa (Other); Bill and Melinda Gates Foundation (Other); Wits Health Consortium (Pty) Ltd (Other); University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ChAdOx1 nCoV-19_ZA_phI/II v4.1
Record Dates: First submitted 2020-06-15; First posted 2020-06-23 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — ChAdOx1 nCoV-19; Saline Solution

STUDY DESIGN:
Intervention Model Description: Four groups will be enrolled to receive either one or two doses of investigational vaccine or placebo. Follow up intensity and blood draws differ between groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded, placebo controlled. Pharmacist and vaccine administrators will be unblinded only. DSMB will be unblinded if required to assess safety signal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group 1- IP (Experimental): Participants (HIV-negative) will receive two doses of 5-7.5x10^10 vp ChAdOx1 nCoV-19 vaccine in deltoid of non-dominant arm, 28 days apart. Participants, investigators and outcome assessors will be blinded to intervention. Participants will have 11 routine visits over a 12 month period.
  Interventions: Biological: ChAdOx1 nCoV-19
- Group 1- placebo (Placebo Comparator): Participants (HIV-negative) will receive two doses of Normal saline (0.9%) in deltoid of non-dominant arm, 28 days apart. Participants, investigators and outcome assessors will be blinded to intervention. Participants will have 11 routine visits over a 12 month period.
  Interventions: Biological: Normal saline 0.9%
- Group 2a- IP (Experimental): Participants (HIV-negative) will receive two doses of 5-7.5x10^10 vp ChAdOx1 nCoV-19 vaccine in deltoid of non-dominant arm, 28 days apart. Participants, investigators and outcome assessors will be blinded to intervention. Participants will have 7 (1-dose) or 9 (2 doses) routine visits over a 12 month period.
  Interventions: Biological: ChAdOx1 nCoV-19
- Group 2a- placebo (Placebo Comparator): Participants (HIV-negative) will receive two doses of placebo in deltoid of non-dominant arm, 28 days apart. Participants, investigators and outcome assessors will be blinded to intervention. Participants will have 7 (1-dose) or 9 (2 doses) routine visits over a 12 month period.
  Interventions: Biological: Normal saline 0.9%
- Group 2b- IP (Experimental): Participants will receive two doses of 5-7.5x10^10 vp ChAdOx1 nCoV-19 vaccine in deltoid of non-dominant arm, 28 days apart. Participants, investigators and outcome assessors will be blinded to intervention. Participants will have 5 (1-dose) or 6 (2 doses) routine visits over a 12 month period.
  Interventions: Biological: ChAdOx1 nCoV-19
- Group 2b- placebo (Placebo Comparator): Participants will receive two doses of placebo in deltoid of non-dominant arm, 28 days apart. Participants, investigators and outcome assessors will be blinded to intervention. Participants will have 5 (1-dose) or 6 (2 doses) routine visits over a 12 month period.
  Interventions: Biological: Normal saline 0.9%
- Group 3- IP (Experimental): Participants (HIV-positive) will receive two doses of 5-7.5x10^10 vp ChAdOx1 nCoV-19 vaccine in deltoid of non-dominant arm, 28 days apart. Participants, investigators and outcome assessors will be blinded to intervention. Participants will have 11 routine visits over a 12 month period.
  Interventions: Biological: ChAdOx1 nCoV-19
- Group 3- placebo (Placebo Comparator): Participants (HIV-positive) will receive two doses of placebo in deltoid of non-dominant arm, 28 days apart. Participants, investigators and outcome assessors will be blinded to intervention. Participants will have 11 routine visits over a 12 month period.
  Interventions: Biological: Normal saline 0.9%

INTERVENTIONS:
Biological: ChAdOx1 nCoV-19 — Dose of 5-7.5x10^10vp of ChAdOx1 nCoV-19
  Arms: Group 1- IP; Group 2a- IP; Group 2b- IP; Group 3- IP
Biological: Normal saline 0.9% — Normal saline 0.9% as placebo
  Arms: Group 1- placebo; Group 2a- placebo; Group 2b- placebo; Group 3- placebo

SUMMARY:
A Phase I/II, double-blinded, placebo-controlled, individually randomized trial to assess safety, immunogenicity and efficacy of the candidate Coronavirus disease (COVID-19) vaccine ChAdOx1 nCoV-19 in adults aged 18-65 years living with and without HIV in South Africa. The vaccine or placebo will be administered via an intramuscular injection into the deltoid muscle of the non-dominant arm.

DETAILED DESCRIPTION:
A total of 2070 participants will be enrolled into the trial; 1970 HIV-uninfected and 100 people living with HIV. There will be 4 trial groups, group 1 (n=50; intensive safety & immunogenicity cohort, HIV negative), group 2a (n=250; safety, intense immunogenicity & efficacy), group 2b (n=1650; safety, immunogenicity & vaccine efficacy) and group 3 (n=100, intensive safety & immunogenicity cohort, HIV positive).

Participants will be followed up for 12 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-65 years.
* Documented result of not being infected with HIV (including screening by a rapid HIV antibody test) within two weeks of randomization into the study for Group-1 and Group-2 participants only.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow investigators review available medical records, and review all medical and laboratory records if participant is admitted to hospital with respiratory tract infection suspected or confirmed to be COVID-19.
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening (within 14 days of randomization) or vaccination.
* For Group-3 only (i.e. HIV-infected), need to have been on anti-retroviral treatment for at least three months and HIV-1 viral load is <1,000 copies/ml within two weeks of randomization.
* Agreement to refrain from blood donation during the course of the study.
* Provide written informed consent.

Exclusion Criteria:

* Planned receipt of any vaccine other (licensed or investigational) than the study intervention within 30 days before and after each study vaccination.
* Use of any unproven registered and unregistered treatments for COVID-19.
* Prior receipt of an investigational or licensed vaccine likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccines, any coronavirus vaccines).
* Administration of immunoglobulins and/ or any blood products within the three months preceding the planned administration of the vaccine candidate.
* HBSAg positivity on the screening sample.
* Grade 2 or higher level of abnormality for FBC, U&E or LFT based on DAIDS Grading Criteria (Version 2.1, July 2017)
* History of allergic disease or reactions likely to be exacerbated by any component of the ChAdOx1 nCoV-19 vaccine.
* Any history of hereditary angioedema or idiopathic angioedema.
* Any history of anaphylaxis in relation to vaccination.
* Pregnancy, lactation or willingness/intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition likely to affect participation in the study.
* Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture.
* Any other serious chronic illness requiring hospital specialist supervision.
* Chronic respiratory diseases, including asthma
* Chronic cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness
* Seriously overweight (BMI ≥ 40 Kg/m2)
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrollment.
* Any clinically significant abnormal finding on screening urinalysis.
* Any other significant disease, disorder or finding which may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study or impair interpretation of the study data.
* History of laboratory confirmed COVID-19 illness or known contact with a person that was infected with SARS-COV-2.
* New onset of fever or a cough or shortness of breath in the 30 days preceding screening and/or enrollment
* Travel history to any other country with widespread epidemic since January 2020
* In addition to above, Group 1 & 2 participants need to fulfill the following exclusion criteria: Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent severe infections and chronic use (more than 14 days) immunosuppressant medication within the past 6 months ( topical steroids are allowed).
* Any confirmed or suspected immunosuppressive or immunodeficient state (except HIV infection for Group-3), asplenia, recurrent severe infections and chronic use (more than 14 days) immunosuppressant medication within the past 6 months (topical steroids are allowed).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2130 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence of adverse events (intervention-related and intervention-unrelated) in HIV-negative adults aged 18-65 year receiving candidate ChAdOx1 nCoV-19 vaccine or placebo (safety) | Up to 12 months post enrollment
  Number of solicited local and systemic reactogenicity signs and symptoms for 7 days following vaccination, and unsolicited adverse events for 28 days following vaccination.
  Assess occurrence of disease enhancement episodes and serious adverse events in year post vaccination
Determine if there is a reduction of severe and non-severe COVID-19 disease in HIV-negative adults who receive candidate vaccine ChAdOx1 nCoV-19 compared to placebo recipients (efficacy) | Up to 12 months post enrollment
  Virologically-confirmed COVID-19 clinical disease will be defined as an acute respiratory illness that is clinically consistent with COVID-19 disease, AND SARS-CoV-2 RT-PCR positivity.
Assess the incidence of adverse events (intervention-related and intervention-unrelated) in HIV-positive adults aged 18-65 year receiving candidate ChAdOx1 nCoV-19 vaccine or placebo (safety) | Up to 12 months post enrollment
  Number of solicited local and systemic reactogenicity signs and symptoms for 7 days following vaccination, and unsolicited adverse events for 28 days following vaccination.
  Assess occurrence of disease enhancement episodes and serious adverse events in year post vaccination
Assess cellular Immunogenicity of ChAdOx1 nCoV-19 in people living with HIV (immunogenicity) | Up to 12 months post enrollment
  Assessing the Interferon-gamma (IFN-γ) enzyme- linked immunospot (ELISpot) responses to SARS-CoV-2 spike protein and Th1 and Th2 cytokine response profile at 3-4 days after vaccination
Assess humoral immunogenicity of ChAdOx1 nCoV-19 in people living with HIV | Up to 12 months post enrollment
  Assessing Enzyme-linked immunosorbent assay (ELISA) or fluorescence based micro-bead immunosorbent assay on luminex platform to quantify antibodies against SARS-CoV-2 spike protein (seroconversion rates) and Virus neutralising antibody (NAb) assays against live and/or pseudotyped SARS-CoV-2 virus

SECONDARY OUTCOMES:
Assess humoral Immunogenicity of ChAdOx1 nCoV-19 in HIV-negative adults (immunogenicity) | Up to 12 months post enrollment
  Assessing Enzyme-linked immunosorbent assay (ELISA) or fluorescence based micro-bead immunosorbent assay on luminex platform to quantify antibodies against SARS-CoV-2 spike protein (seroconversion rates) and Virus neutralising antibody (NAb) assays against live and/or pseudotyped SARS-CoV-2 virus
Assess cellular Immunogenicity of ChAdOx1 nCoV-19 in HIV-negative adults (immunogenicity) | Up to 12 months post enrollment
  Assessing the Interferon-gamma (IFN-γ) enzyme- linked immunospot (ELISpot) responses to SARS-CoV-2 spike protein and Th1 and Th2 cytokine response profile at 3-4 days after vaccination

OTHER OUTCOMES:
Assess Fc effector functionality in participants who receive ChAdOx1 nCoV-19 vaccine or placebo | Up to 12 months post enrollment
  Cellular Fc effector functionality assays to measure the ability of vaccine elicited antibodies to mediate cellular cytotoxicity, complement deposition, and phagocytosis.
Assess B cell responses to SARS-CoV-2 spike trimer and/or the receptor binding domain in participants who receive ChAdOx1 nCoV-19 vaccine or placebo | Up to 12 months post enrollment
  Flow cytometric sorting of plasmablasts and memory B cells to using spike and receptor binding domain "baits" to isolate SARS-CoV-2 specific B cells, sequence their immunoglobulin genes and define their epitope specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, MD, PhD, Principal Investigator — University of Witwatersrand, South Africa
Locations (7):
- South Africa (7):
  - PHRU Kliptown, Johannesburg, Gauteng
  - Soweto Clinical Trials Centre, Johannesburg, Gauteng
  - Wits RHI Shandukani Research Centre, Johannesburg, Gauteng
  - Setshaba Research Centre (SRC), Soshanguve, Gauteng
  - Chris Hani Baragwanath Academic Hospital - DST/NRF VPD RMPRU, Soweto, Gauteng
  - FAMCRU, Cape Town, Western Cape
  - Groote Schuur hospital, Lung infection and immunity unit, UCT, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
The data accumulated from this study will be stored at RMPRU/ Wits. In collaboration with UK collaborators, we aim to make the data available, within one year of completion of the study to any investigators who wish to use the data to address any specific questions not directly addressed under the study objectives and which the data would lend itself to.
  De-identified data will be shared. Related trial documents will be available (protocol, ICFs, statistical analysis plan)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within 1 year of trial completion
Access Criteria: Any investigators who wish to use the data to address any specific questions not directly addressed under the study objectives and which the data would lend itself to.

REFERENCES:
- [Derived] Koen AL, Izu A, Baillie V, Kwatra G, Cutland CL, Fairlie L, Padayachee SD, Dheda K, Barnabas SL, Bhorat QE, Briner C, Ahmed K, Bhikha S, Bhiman JN, du Plessis J, Esmail A, Horne E, Hwa SH, Oommen-Jose A, Lambe T, Laubscher M, Malahleha M, Benade G, McKenzie S, Oelofse S, Patel F, Pillay S, Rhead S, Rodel H, Taoushanis C, Tegally H, Thombrayil A, Villafana TL, Gilbert S, Pollard AJ, Madhi SA. Efficacy of primary series AZD1222 (ChAdOx1 nCoV-19) vaccination against SARS-CoV-2 variants of concern: Final analysis of a randomized, placebo-controlled, phase 1b/2 study in South African adults (COV005). Vaccine. 2023 May 26;41(23):3486-3492. doi: 10.1016/j.vaccine.2023.04.058. Epub 2023 Apr 27. PMID 37149443
- [Derived] Smith M, Kwatra G, Izu A, Nel A, Cutland C, Ahmed K, Baillie V, Barnabas S, Bhorat Q, Briner C, Lazarus E, Dheda K, Fairlie L, Koen A, Madhi S, Blackburn JM. Longitudinal IgA and IgG Response, and ACE2 Binding Blockade, to Full-Length SARS-CoV-2 Spike Protein Variants in a Population of Black PLWH Vaccinated with ChAdOx1 nCoV-19. Viruses. 2023 Feb 6;15(2):448. doi: 10.3390/v15020448. PMID 36851662
- [Derived] Madhi SA, Kwatra G, Richardson SI, Koen AL, Baillie V, Cutland CL, Fairlie L, Padayachee SD, Dheda K, Barnabas SL, Bhorat QE, Briner C, Ahmed K, Aley PK, Bhikha S, Bhorat AE, Esmail A, Horne E, Kaldine H, Mukendi CK, Madzorera VS, Manamela NP, Masilela M, Hermanus ST, Motlou T, Mzindle N, Oelofse S, Patel F, Rhead S, Rossouw L, Taoushanis C, van Eck S, Lambe T, Gilbert SC, Pollard AJ, Moore PL, Izu A. Durability of ChAdOx1 nCoV-19 (AZD1222) vaccine and hybrid humoral immunity against variants including omicron BA.1 and BA.4 6 months after vaccination (COV005): a post-hoc analysis of a randomised, phase 1b-2a trial. Lancet Infect Dis. 2023 Mar;23(3):295-306. doi: 10.1016/S1473-3099(22)00596-5. Epub 2022 Oct 20. PMID 36273491
- [Derived] Madhi SA, Koen AL, Izu A, Fairlie L, Cutland CL, Baillie V, Padayachee SD, Dheda K, Barnabas SL, Bhorat QE, Briner C, Aley PK, Bhikha S, Hermanus T, Horne E, Jose A, Kgagudi P, Lambe T, Masenya M, Masilela M, Mkhize N, Moultrie A, Mukendi CK, Moyo-Gwete T, Nana AJ, Nzimande A, Patel F, Rhead S, Taoushanis C, Thombrayil A, van Eck S, Voysey M, Villafana TL, Vekemans J, Gilbert SC, Pollard AJ, Moore PL, Kwatra G; Wits VIDA COVID team. Safety and immunogenicity of the ChAdOx1 nCoV-19 (AZD1222) vaccine against SARS-CoV-2 in people living with and without HIV in South Africa: an interim analysis of a randomised, double-blind, placebo-controlled, phase 1B/2A trial. Lancet HIV. 2021 Sep;8(9):e568-e580. doi: 10.1016/S2352-3018(21)00157-0. Epub 2021 Aug 17. PMID 34416193
- [Derived] Madhi SA, Baillie V, Cutland CL, Voysey M, Koen AL, Fairlie L, Padayachee SD, Dheda K, Barnabas SL, Bhorat QE, Briner C, Kwatra G, Ahmed K, Aley P, Bhikha S, Bhiman JN, Bhorat AE, du Plessis J, Esmail A, Groenewald M, Horne E, Hwa SH, Jose A, Lambe T, Laubscher M, Malahleha M, Masenya M, Masilela M, McKenzie S, Molapo K, Moultrie A, Oelofse S, Patel F, Pillay S, Rhead S, Rodel H, Rossouw L, Taoushanis C, Tegally H, Thombrayil A, van Eck S, Wibmer CK, Durham NM, Kelly EJ, Villafana TL, Gilbert S, Pollard AJ, de Oliveira T, Moore PL, Sigal A, Izu A; NGS-SA Group; Wits-VIDA COVID Group. Efficacy of the ChAdOx1 nCoV-19 Covid-19 Vaccine against the B.1.351 Variant. N Engl J Med. 2021 May 20;384(20):1885-1898. doi: 10.1056/NEJMoa2102214. Epub 2021 Mar 16. PMID 33725432
- [Derived] Voysey M, Costa Clemens SA, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Clutterbuck EA, Collins AM, Cutland CL, Darton TC, Dheda K, Dold C, Duncan CJA, Emary KRW, Ewer KJ, Flaxman A, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Galiza E, Goodman AL, Green CM, Green CA, Greenland M, Hill C, Hill HC, Hirsch I, Izu A, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Libri V, Lillie PJ, Marchevsky NG, Marshall RP, Mendes AVA, Milan EP, Minassian AM, McGregor A, Mujadidi YF, Nana A, Padayachee SD, Phillips DJ, Pittella A, Plested E, Pollock KM, Ramasamy MN, Ritchie AJ, Robinson H, Schwarzbold AV, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, White T, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Single-dose administration and the influence of the timing of the booster dose on immunogenicity and efficacy of ChAdOx1 nCoV-19 (AZD1222) vaccine: a pooled analysis of four randomised trials. Lancet. 2021 Mar 6;397(10277):881-891. doi: 10.1016/S0140-6736(21)00432-3. Epub 2021 Feb 19. PMID 33617777
- [Derived] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989